CLINICAL TRIAL: NCT05349838
Title: An Open-Label, Multi-Centre, Randomised, Switch Study to Evaluate the Virological Efficacy Over 96 Weeks Of 2-Drug Therapy With DTG/RPV FDC in Antiretroviral Treatment-Experienced HIV-1 Infected Subjects Virologically Suppressed With Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTIs) Resistance Mutation K103N
Brief Title: Open-Label Multi-Centre Randomised Switch Study to Evaluate Virological Efficacy Over 96Weeks Of 2-Drug Therapy With Dolutegravir(DTG)/Rilpivirine(RPV) Fixed Dose Combination(FDC) in Antiretroviral Treatment-Experienced HIV-1 Infected Subjects Virologically Suppressed With NNRTI Mutation K103N
Acronym: WISARD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NEAT ID Foundation (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEAT 33; 2017-004040-38 (EudraCT Number)
Record Dates: First submitted 2019-05-02; First posted 2022-04-27 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — dolutegravir; Psychotherapy, Multiple

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DTG/RPV FDC Regimen (Experimental): One combined Dolutegravir 50mg /Rilpivirine 25mg FDC tablet taken orally once daily
  Interventions: Drug: Dolutegravir & Rilpivirine 2 drug fixed dose combined therapy
- Continued ART Regimen (Active Comparator): Patients will continue the current boosted PI regimen (or other antiretroviral combination) for 48 weeks. Patients will then be switched to one combined Dolutegravir/Rilpivirine FDC tablet taken orally once daily for 48 weeks.
  Interventions: Drug: Dolutegravir & Rilpivirine 2 drug fixed dose combined therapy

INTERVENTIONS:
Drug: Dolutegravir & Rilpivirine 2 drug fixed dose combined therapy — Daily oral tablet
  Other Names: Boosted protease inhibitors or other ARV regimen

SUMMARY:
HIV-1 infected subjects that experience virological failure while on non nucleoside reverse-transcriptase inhibitors (NNRTIs), including those with the K103N mutation, are usually switched to a boosted Protease Inhibitor (PI)-based regimen or other antiretroviral (ARV) combinations. The same is true for subjects who need to start antiretroviral therapy and have acquired virus that is already resistant to antiretrovirals. These "second line" combinations are often associated with numerous issues that can have a potential impact on the quality of life (QoL) of these patients. Therefore a simpler and better tolerated alternative second line treatment option would be a useful tool for the clinical management of these patients.

The aim of this study is to assess the efficacy and tolerability of a dual combined therapy of Dolutegravir (DTG) 50 mg Once Daily (OD) + Rilpivirine (RPV) 25 mg OD in virologically suppressed participants with previous virological failure with NNRTIs and having the clinically significant mutation K103N. The secondary objective of the study is to assess whether a simplification of the treatment in terms of pill burden, long term metabolic toxicity and potential for drug interactions improves the QOL of the participants. The study will also evaluate DTG & RPV concentrations in the blood plus changes in cell associated virus.

In order to compare the first line treatment (boosted PI and/or other antiretroviral combinations) and the DTG+RPV combination, two thirds of study participants will be switched to DTG+RPV immediately and receive DTG+RPV for 96 weeks. The other third will be switched after 48 weeks of continuing on their first line treatment and receive DTG+RPV for 48 weeks. All participants will then be followed up for a further 30 days. Participants will be recruited from sites across Europe, and randomised onto either arm of the study. After randomisation, participants will attend approximately 10 visits over the course of two years.

ELIGIBILITY:
Inclusion criteria

Patient volunteers who meet all of the following criteria are eligible for this trial:

1. Is male or female aged 18 years or over.
2. Has documented HIV-1 infection
3. Is capable of giving informed consent
4. Is willing to comply with the protocol requirements
5. Virologically suppressed (plasma HIV-RNA <50 copies/mL for >24 weeks) and on a stable regimen.
6. Subjects are required to have a history of the K103N mutation (acquired or selected). Subjects who at any time have had the mutations 100I, 101E/P, 106A/M, 138K/G/Q, 181C/I/V, 188L, 190A/S/E/Q, 230L mutations are to be excluded. Other NNRTI region variants can be included. All PI and NRTI mutations are acceptable. Study sites may ask the coordinating centre for advice as required.
7. Subjects must have never failed INSTI (2 x VL >200 >2 weeks apart) but current regimen can include Integrase Strand Transfer Inhibitor(INSTI).
8. A female, may be eligible to enter and participate in the study if she:

   a. is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea without an alternative medical cause and ≥ 45 years of age) A high follicle stimulating hormone (FSH) level consistent with postmenopausal status may be used to confirm a post- menopausal state in women who are not using hormonal contraception) or hormonal replacement therapy at the discretion of the Principal Investigator. However, in the absence of 12 months of amenorrhea, a single FSH measurement alone is insufficient.

   OR physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,

   OR is of child-bearing potential with a negative pregnancy test at Screening (& baseline visit) and agrees to use one of the following methods of contraception to avoid pregnancy:

   True abstinence from penile-vaginal intercourse from 2 weeks prior to administration of IP, throughout the study, and for at least 2 weeks after discontinuation of all study medications (When this is in line with the preferred and usual lifestyle of the subject.) (Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), and withdrawal are not acceptable methods of contraception.

   Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion, see Appendix 3 for an example listing of approved IUDs).

   Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject;

   Approved hormonal contraception (see appendix 4 for a listing of examples of approved hormonal contraception);

   Any other method with published data showing that the expected failure rate is <1% per year.

   Any contraceptive method must be used consistently and for at least 2 weeks after discontinuation of Investigational Product (IP)
9. If a heterosexually active male, he is using effective birth control methods and is willing to continue practising these birth control methods during the trial and until follow-up visit
10. Subjects currently receiving DTG or RPV, but not both, can be included.

Exclusion criteria

Patients meeting 1 or more of the following criteria cannot be selected:

1. Infected with HIV-2
2. Detectable HIV-1 RNA at screening (HIV-1 RNA measurement >=50 c/mL).
3. Subjects requiring regular dosing doing with H2 or PPI antacid medications or a history of achlorhidria or drug known to interact with RPV or DTG.
4. Use of medications which are associated with Torsades de Pointes
5. Corrected QT interval (QTc [Bazett]) >450 milliseconds or QTc (Bazett) >480 milliseconds for participants with bundle branch block. The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB).
6. Unstable health conditions (i.e. opportunistic infections, cancers, unstable liver disease etc).
7. Any evidence of an active Centers for Disease Control and Prevention Category C disease. Exceptions include cutaneous Kaposi's sarcoma not requiring systemic therapy and historic CD4+ lymphocyte counts of <200 cells/millimeter3.
8. History or presence of allergy to the study drugs or their components or drugs of their class;
9. Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the Study medical monitor for inclusion of the subject prior to randomization;
10. Any pre-existing physical or mental condition which, in the opinion of the Investigator, may interfere with the subject's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participants. Subjects considered to pose a significant risk of suicide should be excluded.
11. Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the subject unable to take oral medication;
12. Using any concomitant therapy disallowed as per the reference safety information and product labelling for the study drugs. Specifically, co-administration with the following medicinal products is not allowed:

    * dofetilide or pilsicainide;
    * fampridine (also known as dalfampridine);
    * carbamazepine, oxcarbazepine, phenobarbital, phenytoin;
    * rifampicin, rifapentine;
    * proton pump inhibitors, such as omeprazole, esomeprazole, lansoprazole, pantoprazole, rabeprazole; - systemic dexamethasone, except as a single dose treatment;
    * St John's wort (Hypericum perforatum).
13. Has acute viral hepatitis including, but not limited to, A, B, or C
14. Active hepatitis B/ Hep B non-immune subjects who have failed vaccination (antibody concentration < 10 international units). (If local practice does not include vaccination of low risk patients, then the patients without HBsAb are not excluded - this must be clearly documented in the medical records and eCRF). (Note: subjects can be re screened if they receive vaccination and subsequently meet eligibility criteria)
15. Evidence of Hepatitis B virus (HBV) infection based on the results of testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), and Hepatitis B surface antibody (HBsAb) as follows: Participants positive for HBsAg are excluded; Participants positive for anti-HBc (negative HBsAg status) and negative for HBsAb are excluded. (if local practice does not include vaccination of low risk patients, then the patients without HBsAb are not excluded - this must be clearly documented in the medical records and eCRF. Note: Subject positive for anti-HBc (negative HBsAg status) and positive for HBsAb are immune to HBV and are not excluded.
16. Participants with an anticipated need for any Hepatitis C virus (HCV) therapy during the Early Switch Phase and for interferon-based therapy for HCV throughout the entire study period.
17. Any investigational drug within 30 days prior to the trial drug administration
18. Any evidence of viral resistance different to the one described in the inclusion criteria i.e. not meeting inclusion criteria or having different mutation at K103.
19. Dialysis or renal insufficiency (creatinine clearance < 50ml/min)
20. History of decompensated liver disease (Alanine aminotransferase (ALT) ≥ 5 times the upper limit of normal (ULN), OR ALT ≥3xULN and bilirubin ≥1.5xULN (with >35% direct bilirubin)
21. Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
22. Subjects with severe hepatic impairment (Class C) as determined by Child-Pugh classification (see appendix 4)
23. Opportunistic infection within 4 weeks prior to first dose of DTG plus RPV.
24. Clinical decision that a switch of antiretroviral therapy should be immediate
25. Screening blood result with any grade 3/4 toxicity according to Division of AIDS (DAIDS) grading scale, except: asymptomatic grade 3 glucose, amylase or lipid elevation or asymptomatic grade 4 triglyceride elevation (re-test allowed). or unconjugated hyperbilirubinaemia due to atanazavir exposure.
26. Any condition (including illicit drug use or alcohol abuse) or laboratory results which, in the investigator's opinion, interfere with assessments or completion of the trial.
27. Women planning pregnancy or who are pregnant or breast feeding. (NB: See section 6.12 Withdrawal Criteria for guidance if pregnancy does occur).
28. Females of childbearing potential and males must be willing to use a highly effective (acceptable effective contraceptive measures are only acceptable for IMP's with unlikely human teratogenicity / fetotoxicity in early pregnancy) method of contraception (hormonal method of birth control; true abstinence). Contraceptive methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods (see Appendix 4). Such methods include:

    * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral intravaginal transdermal
    * progesteron-only hormonal contraception associated with inhibition of ovulation oral injectable implantable
    * Intrauterine device (IUD)
    * Intrauterine hormone-releasing system ( IUS)
    * bilateral tubal occlusion
    * vasectomized partner
    * true sexual abstinence

    (NB: See section 6.12 Withdrawal Criteria for guidance if pregnancy does occur).
29. Hypersensitivity to the active substances or to any of the excipients listed below: List of excipients Tablet core • Mannitol (E421) • Magnesium stearate • Microcrystalline cellulose • Povidone (K29/32) • Sodium starch glycolate • Sodium stearyl fumarate • Lactose monohydrate • Croscarmellose sodium • Povidone (K30) • Polysorbate 20 • Silicified microcrystalline cellulose Tablet coating • Polyvinyl alcohol- part hydrolysed • Titanium dioxide (E171) • Macrogol • Talc • Iron oxide yellow (E172) Iron oxide red (E172)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- Belgium (2):
  - Institute of Tropical Medecine, Antwerp
  - St Pierre University Hospital, Brussels
- France (3):
  - CHU Hotel Dieu, Nantes
  - Hospital Saint Louis, Paris
  - Pitié-salpêtrière Hospital, Paris
- Germany (4):
  - University Bonn, Bonn
  - University Essen, Essen
  - Frankfurt University Hospital, Frankfurt
  - ICH Study Center, Hamburg, Hamburg
- Italy (5):
  - AAST delgi spedali civili di Brescia, Brescia
  - ASST FBF SACCO- I Division of Infectious Diseases 1, Milan
  - ASST FBF SACCO- I Division of Infectious Diseases 3, Milan
  - I.R.C.C.S San Raffaele Hospital, Milan
  - ASST GOM Niguarda Milano, Dep. Infectious Disease, Milan
- Spain (6):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Herbo, Barcelona
  - Infectious Diseases Unit Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario La Paz, Madrid, Madrid
- United Kingdom (9):
  - Brighton & Sussex University NHS Trust, Brighton
  - North Bristol NHS Trust, Southmead Hospital, Bristol
  - Chelsea & Westminster Hospital, London
  - Kings College Hospital London, London
  - Mortimer Market Centre, London
  - Queen Elizabeth Hospital, London
  - Royal Free London NHS Foundation Trust, London
  - St Marys Hospital, London
  - The Royal London Hospital, London

REFERENCES:
- [Derived] Moyle G, Assoumou L, de Castro N, Post FA, Curran A, Rusconi S, De Wit S, Stephan C, Raffi F, Johnson M, Masia M, Vera J, Jones B, Grove R, Fletcher C, Duffy A, Morris K, Pozniak A; NEAT ID Foundation and the WISARD study group. Switching to dolutegravir plus rilpivirine versus maintaining current antiretroviral therapy regimen in virologically suppressed people with HIV-1 and the Lys103Asn (K103N) mutation: 48-week results from a randomised, open-label pilot clinical trial. Lancet HIV. 2024 Mar;11(3):e156-e166. doi: 10.1016/S2352-3018(23)00292-8. PMID 38417976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 32 medical centres across Europe. The first participant was enrolled in November 2018 and the last participant was enrolled in December 2020.
Pre-assignment Details: Of 176 participants that were screened for the study, 140 met eligibility criteria and were randomised to the study.
Period: Overall Study
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Started | 95 | 45
Per-protocol Population at Week 48 | 87 | 40
Completed | 83 | 36
Not Completed | 12 | 9
Not completed — Virological Failure | 1 | 2
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Other reasons | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen | Total
Number analyzed (Participants) | 95 | 45 | 140
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [44 to 58] | 53 [47 to 56] | 52 [46 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 79 | 35 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity N(%): White caucasian | 69 | 29 | 98
  Ethnicity N(%): White mixed | 2 | 1 | 3
  Ethnicity N(%): Asian | 4 | 0 | 4
  Ethnicity N(%): Black | 7 | 7 | 14
  Ethnicity N(%): African | 3 | 3 | 6
  Ethnicity N(%): Caribbean | 1 | 1 | 2
  Ethnicity N(%): Other | 9 | 4 | 13
Region of Enrollment [Number; unit: participants]
  Belgium | 6 | 3 | 9
  United Kingdom | 36 | 16 | 52
  Italy | 7 | 3 | 10
  France | 23 | 13 | 36
  Germany | 8 | 2 | 10
  Spain | 15 | 7 | 22
  Ireland | 0 | 1 | 1
Body Mass Index (BMI) (kg/m^2) [Median (Inter-Quartile Range); unit: kg/m^2] | 24.3 [22 to 28] | 26.4 [24 to 29] | 25.1 [23 to 28]
Drinks alchohol [Count of Participants; unit: Participants] | 52 | 25 | 77
Current smoker [Count of Participants; unit: Participants] | 34 | 12 | 46
Uses recreational drugs [Count of Participants; unit: Participants] | 15 | 7 | 22
Hypertension [Count of Participants; unit: Participants] | 14 | 8 | 22
Diabetes [Count of Participants; unit: Participants] | 6 | 4 | 10
Hepatitis C IgG antibodies [Count of Participants; unit: Participants] | 9 | 3 | 12
Hepatitis B core antibodies [Count of Participants; unit: Participants] | 28 | 17 | 45
Hepatitis B surface antibodies [Count of Participants; unit: Participants] | 80 | 36 | 116
HIV Information [Median (Inter-Quartile Range); unit: years]
  Years since HIV diagnosis | 17.1 [7.3 to 26.3] | 22.4 [13.1 to 26.5] | 19.7 [8.8 to 26.4]
  Years on ART | 16 [6.3 to 23] | 17.7 [10.5 to 23] | 16.5 [7.3 to 23]
ART at enrolment [Count of Participants; unit: Participants]
  Nucleoside Reverse Transcriptase Inhibitor (NRTI) regimen | 72 | 36 | 108
  Tenofovir-DF (TDF) / Emtrictabine | 25 | 7 | 32
  Tenofovir-AF (TDF) / Emtrictabine | 22 | 15 | 37
  Abcavir/Lamivudine | 17 | 8 | 25
  Other | 8 | 5 | 13
  PI regimen | 60 | 27 | 87
  Darunavir | 50 | 22 | 72
  Atazanavir | 8 | 5 | 13
  Lopinavir | 1 | 0 | 1
  Amprenavir | 1 | 0 | 1
  Integrase Strand Transfer Inhibitor (INSTI) regimen | 46 | 21 | 67
  Raltegravir | 16 | 7 | 23
  Dolutegravir | 20 | 8 | 28
  Bictegravir | 3 | 1 | 4
  Elvitegravir | 7 | 5 | 12
  Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI) regimen | 7 | 6 | 13
  Etravirine | 6 | 4 | 10
  Rilpivirine | 1 | 2 | 3
History of HIV-1 resistance mutations [Median (Inter-Quartile Range); unit: Number of mutations]
  Total number of drug resistance mutations according to IAS 2019 | 3 [1 to 6] | 4 [1 to 7] | 3 [1 to 6]
  Total number of NRTI drug resistance mutations according to IAS 2019 | 1 [0 to 2] | 1 [0 to 3] | 1 [0 to 2]
  Total number of NNRTI drug resistance mutations according to IAS 2019 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Total number of PI drug resistance mutations according to IAS 2019 | 0 [0 to 2] | 1 [0 to 3] | 1 [0 to 3]
Frequency of other Nucleoside Non-nucleoside reverse transcriptase inhibitors resistance mutations [Count of Participants; unit: Participants]
  Leu100Ile | 0 | 0 | 0
  Lys101Glu/Pro | 0 | 0 | 0
  Val106Ala/Ile/Met/Thr | 1 | 3 | 4
  Val108Ile | 7 | 4 | 11
  Glu138Ala/Gly/Lys/Gln/Arg | 0 | 0 | 0
  Val179Asp/Phe/Thr/Leu | 2 | 1 | 3
  Tyr181Cys/Ile/Val | 0 | 0 | 0
  Tyr188Cys/His/Leu | 0 | 0 | 0
  Gly190Ala/Ser/Glu | 0 | 0 | 0
  His221Tyr | 3 | 0 | 3
  Pro225His | 7 | 1 | 8
  Phe227Cys/Leu/Arg | 1 | 0 | 1
  Met230Ile/Leu | 0 | 0 | 0
CD4 CD8 cell count per uL [Median (Inter-Quartile Range); unit: cells/uL] — Population: Data was not collected for one participant
  cells/uL
    CD4+ count: number analyzed (Participants) | 94 | 45 | 139
    CD4+ count | 629 [454 to 800] | 660 [487 to 787] | 650 [464 to 800]
    CD8+ count: number analyzed (Participants) | 94 | 45 | 139
    CD8+ count | 720 [577 to 1015] | 790 [639 to 950] | 753 [578 to 1015]
Cd4 Cd8 % [Median (Inter-Quartile Range); unit: % above versus below 350 cells/μL]
  CD4+ | 33 [26 to 38] | 31 [27 to 38] | 32 [26 to 38]
  CD8+ | 39 [32 to 46] | 39 [33 to 46] | 39 [33 to 46]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With and Without Virological Suppression
Description: Virological Suppression is defined as <50 copies/ml HIV RNA
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 95 | 45
Participants
  HIV RNA < 50 copies/mL | 84 | 40
  HIV RNA >= 50 copies/mL | 3 | 1
  No virologic data at week 48 | 8 | 4

2. Secondary Outcome: Number of Participants With and Without Virological Suppression
Description: Virological Suppression is defined as <50 copies/ml HIV RNA
Time Frame: week 96
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 95 | 45
Participants
  HIV RNA < 50 copies/mL | 80 | 33
  HIV RNA >= 50 copies/mL | 5 | 3
  No virologic data at week 96 | 10 | 9

3. Secondary Outcome: Changes in Blood Cell Counts - Red Blood Cells
Description: red blood cell count evaluation
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Population: Only 93 out of the 95 subjects randomised to the experimental arm (DTG/RPV FDC Regimen) had Red Blood Cell values recorded at baseline. This is the reason the participants analyzed in this category differs from the Participant Flow
Measure: Mean (Standard Error); unit: Red Blood Cells 10^12/L
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 93 | 45
Red Blood Cells 10^12/L
  Change from baseline to week 48 | 0.20 (0.06) | -0.07 (0.09)
  Change from week 48 to week 96 | -0.02 (0.07) | 0.19 (0.10)
  Change from baseline to week 96 | 0.17 (0.09) | 0.12 (0.13)

4. Secondary Outcome: Changes in Blood Cell Counts - White Blood Cells
Description: white blood cell count evaluation
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: White Blood Cells 10^12/L
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 95 | 45
White Blood Cells 10^12/L
  Change from baseline to week 48 | -0.08 (0.26) | -0.06 (0.38)
  Change from week 48 to week 96 | 0.09 (0.27) | -0.03 (0.41)
  Change from baseline to week 96 | 0.01 (0.34) | -0.09 (0.51)

5. Secondary Outcome: Changes in Blood Cell Counts - Platelets
Description: platelet count evaluation
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: Platelets 10^9/L
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 95 | 45
Platelets 10^9/L
  Change from baseline to week 48 | 3.4 (8.2) | -2.6 (12.1)
  Change from week 48 to week 96 | 0.6 (8.6) | 9.3 (13.1)
  Change from baseline to week 96 | 4.0 (11.1) | 6.7 (16.8)

6. Secondary Outcome: Changes in Blood Cell Counts - Haemoglobin
Description: Haemoglobin count evaluation
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 95 | 45
g/dL
  Change from baseline to week 48 | 0.1 (0.2) | 0 (0.3)
  Change from week 48 to week 96 | 0 (0.2) | 0.2 (0.3)
  Change from baseline to week 96 | 0.1 (0.3) | 0.2 (0.4)

7. Secondary Outcome: Change From Baseline in Sodium
Description: Change from baseline in Sodium
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 95 | 45
mmol/L
  Change from baseline to week 48 | 0.3 (0.3) | -0.8 (0.4)
  Change from week 48 to week 96 | -0.5 (0.3) | 0.3 (0.4)
  Change from baseline to week 96 | -0.2 (0.3) | -0.5 (0.5)

8. Secondary Outcome: Changes in Liver Levels - Bilirubin
Description: Liver level evaluation - bilirubin
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 94 | 45
umol/L
  Change from baseline to week 48 | -0.6 (1.4) | -1.9 (2.0)
  Change from week 48 to week 96 | -1.3 (1.4) | -2.2 (2.2)
  Change from baseline to week 96 | -1.9 (1.4) | -4.1 (2.1)

9. Secondary Outcome: Changes in Liver Levels - Alanine Aminotransferase (ALT)
Description: Liver level evaluation - ALT
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: U/L
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 93 | 45
U/L
  Change from baseline to week 48 | 2.4 (3.2) | -0.6 (4.7)
  Change from week 48 to week 96 | -0.7 (3.4) | 1.1 (5.1)
  Change from baseline to week 96 | 1.8 (3.7) | 0.6 (5.6)

10. Secondary Outcome: Changes in Renal Markers - Creatinine Clearance (Estimated Glomerular Filtration Rate(eGFR))
Description: Renal markers evaluation- creatinine clearance (eGFR)
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: eGFR mL/min
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 95 | 44
eGFR mL/min
  Change from baseline to week 48 | -1.7 (2.2) | -1.3 (3.3)
  Change from week 48 to week 96 | -1.2 (2.3) | -3.4 (3.6)
  Change from baseline to week 96 | -2.9 (2.8) | -4.7 (4.2)

11. Secondary Outcome: Change From Baseline in Glucose
Description: Change from baseline in Glucose
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 93 | 43
mmol/L
  Change from baseline to week 48 | -0.15 (0.16) | -0.06 (0.23)
  Change from week 48 to week 96 | 0.09 (0.17) | -0.11 (0.25)
  Change from baseline to week 96 | -0.06 (0.21) | -0.17 (0.31)

12. Secondary Outcome: Changes in Renal Markers - Creatinine
Description: Renal markers evaluation - creatinine
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 95 | 44
umol/L
  Change from baseline to week 48 | 3.0 (2.3) | 0.3 (3.4)
  Change from week 48 to week 96 | 0.3 (2.4) | 5.5 (3.7)
  Change from baseline to week 96 | 3.3 (3.1) | 5.8 (4.7)

13. Secondary Outcome: Changes in Bone Markers - Alkaline Phosphatase
Description: Bone markers evaluation - Alkaline phosphatase
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: U/L
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 94 | 45
U/L
  Change from baseline to week 48 | -5.3 (3.0) | -1.5 (4.3)
  Change from week 48 to week 96 | 3.1 (3.1) | -2.5 (4.7)
  Change from baseline to week 96 | -2.2 (4.0) | -4.0 (6.0)

14. Secondary Outcome: Changes in Fasting Lipids From Baseline - Total Cholesterol
Description: Fasting lipids level evaluation - total cholesterol
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 93 | 45
mmol/L
  Change from baseline to week 48 | -0.09 (0.14) | 0.05 (0.2)
  Change from week 48 to week 96 | 0.02 (0.15) | -0.19 (0.22)
  Change from baseline to week 96 | -0.07 (0.18) | -0.13 (0.27)

15. Secondary Outcome: Changes in Fasting Lipids From Baseline - High Density Lipoprotein (HDL)
Description: Fasting lipids level evaluation - HDL
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 93 | 44
mmol/L
  Change from baseline to week 48 | 0.06 (0.05) | 0.03 (0.07)
  Change from week 48 to week 96 | -0.03 (0.05) | 0.01 (0.08)
  Change from baseline to week 96 | 0.03 (0.06) | 0.04 (0.1)

16. Secondary Outcome: Changes in Quality of Life Health Status Score
Description: Questionnaire (EQ-5D-3L) Mobility, Self-care, Usual activities, Pain/Discomfort and Anxiety/Depression are recorded on 3 point scale (tick boxes), which indicates the severity of problems the participant has with each of these activities. Patients will select No problems, Some problems or Extreme problems/Unable to perform. Patients also report their current Health State on a Scale from 1 to 100 on which the best state you can imagine is marked 100 and the worst state you can imagine is marked 0.
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 93 | 43
score on a scale
  Change from baseline to week 48 | 1.7 (2.9) | 6.3 (4.3)
  Change from week 48 to week 96 | -2.0 (3.0) | -7.2 (4.6)
  Change from baseline to week 96 | -0.3 (3.3) | -0.9 (5.0)

17. Secondary Outcome: Changes in Patient Satisfaction - HIV Treatment Satisfaction Questionnaire (HIVTSQs)
Description: HIV Treatment Satisfaction Questionnaire (HIVTSQs) Answers are recorded on a scale from 0 to 6, with 0 being least satisfied and 6 being most satisfied.
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: Global satisfaction score
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 94 | 45
Global satisfaction score
  Change from baseline to week 48 | 1.6 (0.6) | 0.7 (0.9)
  Change from week 48 to week 96 | 0.2 (0.6) | 0.4 (1.0)
  Change from baseline to week 96 | 1.8 (0.7) | 1.1 (1.1)

18. Secondary Outcome: Number of Participants With Adverse Events - Baseline to Week 48
Description: Adverse Events reports (AEs, SAEs and treatment discontinuation)
Time Frame: Baseline to week 48
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 95 | 45
Participants
  Any Adverse Events (AEs) | 78 | 33
  Grade 1 | 61 | 25
  Grade 2 | 43 | 13
  Grade 3-4 | 7 | 2
  Missing grade | 6 | 1
  Drug related AEs | 22 | 0
  Drug related grade 3-4 AEs | 1 | 0
  AEs leading to study drug interruption | 4 | 0
  SAEs | 4 | 2

19. Secondary Outcome: Number of Drug Drug Interactions
Description: Comparing the drug interaction outcomes between antiretroviral therapy and co-medications before and after the switch by using the www.hiv-druginteractions.org/ website (within the same study arm)
Time Frame: Baseline, week 24, week 48, week 96
Population: Interaction between DTG or RPV and co-medication. For the Continued ART Regimen Group, baseline looks at interaction between ARV treatment at baseline and co-medication and Week 24 is N/A
Measure: Median (Inter-Quartile Range); unit: Number of Drug Interactions
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 90 | 45
Number of Drug Interactions
  Baseline | 1 [0 to 2] | 1 [0 to 3]
  Week 24: number analyzed (Participants) | 88 | 45
  Week 24 | 1 [0 to 2] | NA [NA to NA] — For the Continued ART Regimen Group, drug drug interactions were not assessed at week 24.
  Week 48: number analyzed (Participants) | 86 | 39
  Week 48 | 1 [0 to 2] | 0 [0 to 1]
  Week 96: number analyzed (Participants) | 81 | 38
  Week 96 | 1 [0 to 2] | 0 [0 to 1]

20. Secondary Outcome: Changes in Fasting Lipids From Baseline - Triglycerides
Description: Fasting lipids level evaluation - triglycerides
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 93 | 45
mmol/L
  Change from baseline to week 48 | -0.26 (0.15) | -0.02 (0.22)
  Change from week 48 to week 96 | 0.14 (0.15) | -0.16 (0.23)
  Change from baseline to week 96 | -0.12 (0.18) | -0.18 (0.27)

21. Secondary Outcome: Changes in Fasting Lipids From Baseline - Low Density Lipoprotein (LDL)
Description: Fasting lipids level evaluation - LDL
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 93 | 42
mmol/L
  Change from baseline to week 48 | -0.05 (0.12) | 0 (0.18)
  Change from week 48 to week 96 | 0.02 (0.12) | -0.14 (0.19)
  Change from baseline to week 96 | -0.02 (0.15) | -0.14 (0.23)

22. Secondary Outcome: Changes in Vital Signs From Baseline - Systolic Blood Pressure
Description: Changes in Vital Signs from baseline - Systolic Blood Pressure
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 93 | 45
mmHg
  Change from baseline to week 48 | -1.4 (2.2) | 4.9 (3.3)
  Change from week 48 to week 96 | -0.1 (2.3) | 5.6 (3.6)
  Change from baseline to week 96 | -1.5 (2.7) | 10.5 (4.1)

23. Secondary Outcome: Changes in Vital Signs From Baseline - Diastolic Blood Pressure
Description: Changes in Vital Signs from baseline - Diastolic Blood Pressure
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 95 | 45
mmHg
  Change from baseline to week 48 | 0.2 (1.5) | 3.1 (2.2)
  Change from week 48 to week 96 | -0.7 (1.6) | 0.8 (2.4)
  Change from baseline to week 96 | -0.5 (1.8) | 4.0 (2.7)

24. Secondary Outcome: Changes in Vital Signs From Baseline - Pulse Rate
Description: Changes in Vital Signs from baseline - Pulse rate
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 95 | 45
beats per minute
  Change from baseline to week 48 | 2.1 (1.6) | 2.7 (2.4)
  Change from week 48 to week 96 | -2.5 (1.8) | -1.5 (2.6)
  Change from baseline to week 96 | -0.4 (2.0) | 1.2 (2.9)

25. Secondary Outcome: Changes in Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI measures several different aspects of sleep, with seven component scores and one composite score. The component scores include questions on subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction.
  Each component score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance to sleep. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: Global PSQI score on a scale
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 88 | 40
Global PSQI score on a scale
  Change from baseline to week 48 | -0.1 (0.3) | -0.7 (0.5)
  Change from week 48 to week 96 | 0 (0.3) | -0.5 (0.5)
  Change from baseline to week 96 | -0.1 (0.3) | -1.2 (0.5)

26. Secondary Outcome: Number of Participants With Adverse Events - Week 48 to Week 96
Description: Adverse Events reports (AEs, SAEs and treatment discontinuation)
Time Frame: From Week 48 to week 96
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 87 | 40
Participants
  Any Adverse Events (AEs) | 54 | 28
  Grade 1 | 36 | 18
  Grade 2 | 20 | 12
  Grade 3-4 | 5 | 5
  Missing grade | 7 | 0
  Drug related AEs | 1 | 5
  Drug related grade 3-4 AEs | 0 | 0
  AEs leading to study drug interruption | 1 | 2
  SAEs | 5 | 1

27. Secondary Outcome: Change From Baseline in CD4
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Population: Change from baseline to week 48, Change from week 48 to week 96; Change from baseline to week 96 in participants in the DTG/RPV FDC Regimen and Continued ART Regimen arms
Measure: Mean (Standard Error); unit: CD4 count cells/mm^3
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 94 | 45
CD4 count cells/mm^3
  Change from baseline to week 48 | -31.7 (34.8) | 9.2 (51)
  Change from week 48 to week 96 | 27.3 (36.3) | -9.8 (55.3)
  Change from baseline to week 96 | -4.4 (47.1) | -0.7 (71.0)

28. Secondary Outcome: Change From Baseline in CD8 Cell Count
Description: Change from baseline to week 48, Change from week 48 to week 96; Change from baseline to week 96 in participants in the DTG/RPV FDC Regimen and Continued ART Regimen arms
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Population: as for outcome 27
Measure: Mean (Standard Error); unit: CD8 cell count: cells/mm^3
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 94 | 45
CD8 cell count: cells/mm^3
  Change from baseline to week 48 | -58.8 (41.3) | 9.7 (60.4)
  Change from week 48 to week 96 | -5.7 (43.2) | -55.8 (66.6)
  Change from baseline to week 96 | -64.5 (53.4) | -46.1 (81.3)

29. Secondary Outcome: Change From Baseline in Body Weight
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Population: Change from baseline to week 48; Change from week 48 to week 96; Change from baseline to week 96 in subjects in DTG/RPV FDC Regimen and Continued ART Regimen arms
Measure: Mean (Standard Error); unit: Body weight, kg
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 95 | 45
Body weight, kg
  Change from baseline to week 48 | 0.7 (2.1) | 1.3 (3.1)
  Change from week 48 to week 96 | 1.7 (2.2) | 1.3 (3.4)
  Change from baseline to week 96 | 2.4 (3.0) | 2.6 (4.5)

30. Secondary Outcome: Change From Baseline in BMI
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Population: Change from baseline to week 48; Change from week 48 to week 96; Change from baseline to week 96 in DTG/RPV FDC Regimen and Continued ART Regimen arms
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 95 | 45
kg/m^2
  Change from baseline to week 48 | 0.3 (0.6) | 0.6 (0.9)
  Change from week 48 to week 96 | 0.5 (0.7) | 0.3 (1.0)
  Change from baseline to week 96 | 0.8 (0.9) | 0.9 (1.3)

31. Other Pre Specified Outcome: Changes in High Sensitivity C-Reactive Protein
Description: High Sensitivity C-Reactive Protein evaluation
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 52 | 24
mg/L
  Change from baseline to week 48 | 0.8 (1.2) | -1.3 (1.8)
  Change from week 48 to week 96 | 0.5 (1.2) | -0.9 (1.9)
  Change from baseline to week 96 | 1.3 (1.4) | -2.2 (2.1)

32. Other Pre Specified Outcome: Changes in CD4/CD8 Ratio
Description: CD4/CD8 evaluation
Time Frame: Changed assessed from baseline to week 48, week 48 to week 96, baseline to week 96
Measure: Mean (Standard Error); unit: ratio
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
Number analyzed (Participants) | 94 | 45
ratio
  Change from Baseline to week 48 | 0.03 (0.06) | 0.02 (0.09)
  Change from week 48 to week 96 | 0.04 (0.06) | 0 (0.1)
  Change from Baseline to week 96 | 0.07 (0.08) | 0.01 (0.13)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from consent until the subject's final study visit (I.e. follow-up visit or end of trial visit). This is on average from the baseline visit (+/- 30 days) until week 96 (+/- 30 days) .
Description: The adverse event reporting period will be from consent until the subject's final study visit (I.e. follow-up visit or end of trial visit). In addition, any untoward event that may occur subsequent to the reporting period that the Investigator assesses as possibly, probably or definitely related to the study drug medication should also be reported as an Adverse Event.
Arm/Group | DTG/RPV FDC Regimen | Continued ART Regimen
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/45
Serious Adverse Events (participants affected / at risk) | 12/95 | 4/45
Other Adverse Events (participants affected / at risk) | 66/95 | 19/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG/RPV FDC Regimen (N=95) | Continued ART Regimen (N=45)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
pachymeningitis (Infections and infestations) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Penile neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0)
pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Legionella infection (Infections and infestations) | 1 (1) | 0 (0)
Atypical mycobacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG/RPV FDC Regimen (N=95) | Continued ART Regimen (N=45)
headache (Nervous system disorders) | 16 (21) | 2 (2)
Insomnia (Psychiatric disorders) | 8 (8) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (7) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 4 (4)
COVID-19 (Infections and infestations) | 9 (9) | 3 (3)
Pyrexia (General disorders) | 5 (5) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Alanine aminotransferase increased (Investigations) | 8 (8) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Urinary tract infection (Infections and infestations) | 6 (7) | 2 (3)
Syphilis (Infections and infestations) | 6 (8) | 2 (2)
Rhinitis (Infections and infestations) | 5 (5) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (12) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Nasopharyngitis (Infections and infestations) | 6 (8) | 5 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Hypertension (Vascular disorders) | 6 (6) | 1 (1)
Blood creatinine increased (Investigations) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT05349838/Prot_001.pdf
  • Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT05349838/SAP_002.pdf